CLINICAL TRIAL: NCT00246766
Title: Qualitative and Quantitative Study of Fetal Movements Using Multichannel Ultrasound Pulsed Doppler in Normal and Pathologic Pregnancy
Brief Title: Study of Fetal Movements Using Multichannel Ultrasound Pulsed Doppler in Normal and Pathologic Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Other Study IDs: CT04/ACTIFOETUS
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Pregnancy; Fetal Distress
Keywords: Maternal's movements recorded by a specific sensor; Parameters of fetal distress (umbilical and cerebral Doppler) and new-born parameters.
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To enable an investigation of fetal movements, the researchers have developed a multichannel ultrasound pulsed Doppler called ACTIFOETUS. This new fetal monitor includes three transducers of four sensors which are placed on three different zones of the mother's abdomen. One of the transducers is aimed at the fetal heart, another at the lower limbs and one transducer at the thorax and the fetal upper limbs to detect heart and body movements. The signals are analysed and processed by software which computes a number of parameters describing the movements.

Ninety pregnant women from 28 weeks gestation will be monitored over a 40 minute period every month or every 2 weeks in case of pathological pregnancy. The final purpose will be to develop a system of home monitoring as an indicator of fetal well-being.

DETAILED DESCRIPTION:
The main objective of the study is to detect quantitative and qualitative disorders of fetal movements from 28 weeks of amenorrhea on a fetus presenting in fetal distress.

The fetal rhythm will be recorded during 24 hours and a correlation between maternal and fetal movements will be studied.

Specific measures:

* The fetal heart rate
* The number and extent of fetal movements

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Pregnancy with singleton
* Woman from 28 weeks of amenorrhea

Exclusion Criteria:

* Fetal malformation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2005-03; Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: François TRANQUART, PR, Principal Investigator — Centre d'Innovation Technologique - CHRU de TOURS
Locations (1):
- University Hospital of TOURS, Tours, France

REFERENCES:
- [Background] Hammacher K, Huter KA, Bokelmann J, Werners PH. Foetal heart frequency and perinatal condition of the foetus and newborn. Gynaecologia. 1968;166(4):349-60. doi: 10.1159/000302346. No abstract available. PMID 5699016
- [Background] Karlsson B, Berson M, Helgason T, Geirsson RT, Pourcelot L. Effects of fetal and maternal breathing on the ultrasonic Doppler signal due to fetal heart movement. Eur J Ultrasound. 2000 Mar;11(1):47-52. doi: 10.1016/s0929-8266(99)00071-3. PMID 10717514
- [Background] Melendez TD, Rayburn WF, Smith CV. Characterization of fetal body movement recorded by the Hewlett-Packard M-1350-A fetal monitor. Am J Obstet Gynecol. 1992 Sep;167(3):700-2. doi: 10.1016/s0002-9378(11)91574-9. PMID 1530026
- [Background] Timor-Tritsch I, Zador I, Hertz RH, Rosen MG. Classification of human fetal movement. Am J Obstet Gynecol. 1976 Sep 1;126(1):70-7. doi: 10.1016/0002-9378(76)90467-1. PMID 961750
- [Background] Shinozuka N, Yamakoshi Y. Measurement of fetal movements using multichannel ultrasound pulsed Doppler: autorecognition of fetal movements by maximum entropy method. Med Biol Eng Comput. 1993 Jul;31 Suppl:S59-66. doi: 10.1007/BF02446651. PMID 8231327
- [Background] Manning FA. Fetal biophysical profile. Obstet Gynecol Clin North Am. 1999 Dec;26(4):557-77, v. doi: 10.1016/s0889-8545(05)70099-1. PMID 10587955